CLINICAL TRIAL: NCT07387640
Title: Synchronized Activation of Core and Pelvic Floor Muscles: A More Effective Strategy for Urinary Incontinence?
Brief Title: Synchronized Core-Pelvic Floor Activation in Urinary Incontinence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Betül Çınar, Lecturer, PhD, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bvubcinar04
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Urinary Incontinence,Stress; Stress Urinary Incontinence; Mixed Incontinence Due to Prolapse of Female Genital Organ; Urinary Incontinence
Keywords: Pelvic floor muscle training; Core stability exercises; Core Muscle Co-activation; Pelvic floor physiotherapy; Surface Electromyography
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor muscle training (Active Comparator): Participants will receive conventional pelvic floor muscle training for 12 weeks, at least three days per week
  Interventions: Other: Conventional Pelvic Floor Muscle Training
- Synchronized Core-Pelvic Floor Muscle Training (Experimental): Participants will receive pelvic floor muscle training combined with co-activation exercises targeting core muscles for 12 weeks at least three days per week
  Interventions: Other: Pelvic Floor and Core Muscle Co-activation Training

INTERVENTIONS:
Other: Conventional Pelvic Floor Muscle Training — Participants will receive conventional pelvic floor muscle training based on standardized pelvic floor physiotherapy principles. Exercises will be performed for 12 weeks, at least three days per week, including one supervised session and two home-based sessions.
  Arms: Pelvic floor muscle training
Other: Pelvic Floor and Core Muscle Co-activation Training — Participants will receive pelvic floor muscle training combined with co-activation exercises targeting core muscles. The program will be conducted for 12 weeks with the same frequency and supervision structure as the control group.
  Arms: Synchronized Core-Pelvic Floor Muscle Training

SUMMARY:
This study aims to investigate whether co-activation of the pelvic floor and core muscles improves treatment outcomes in individuals with urinary incontinence. Participants diagnosed with stress, or mixed urinary incontinence will undergo a 12-week pelvic floor physiotherapy program, with or without additional core muscle co-activation exercises. Changes in urinary incontinence severity, pelvic floor muscle function, core muscle activation, and quality of life will be evaluated.

DETAILED DESCRIPTION:
Urinary incontinence is a prevalent condition that negatively affects quality of life and functional independence. Pelvic floor muscle training (PFMT) is recommended as a first-line conservative treatment. Recent evidence suggests that coordinated activation of the pelvic floor muscles with core muscles, including the transversus abdominis and multifidus, may enhance treatment effectiveness.

This randomized controlled study will include women aged 18-65 years diagnosed with stress or mixed urinary incontinence. Eligible participants will be randomly allocated to one of two groups: a conventional pelvic floor muscle training group (control group) or a pelvic floor muscle training plus core muscle co-activation group (intervention group).

Both groups will participate in a 12-week exercise program performed at least three days per week, including one supervised session and two home-based sessions weekly. Outcome measures will be assessed at baseline and after completion of the intervention. Primary outcomes include urinary incontinence severity, while secondary outcomes include pelvic floor muscle function, core muscle activation assessed by surface electromyography, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Diagnosed with stress, urge, or mixed urinary incontinence
* Pelvic floor muscle strength grade ≥ 3 according to the Modified Oxford Scale
* At least one episode of urinary leakage within the last month

Exclusion Criteria:

* Pregnancy
* Childbirth within the previous 6 weeks
* Severe pelvic organ prolapse
* Active vaginal or urinary tract infection
* Presence of neurological or psychiatric disorders
* Malignancy
* Inability to cooperate with assessments or interventions

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Being women
Enrollment: 50 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire | 12 weeks
  This is a brief patient-reported questionnaire used to assess the frequency, severity, and impact of urinary incontinence on quality of life.
  Minimum Score: 0
  Maximum Score: 21
  Interpretation: Higher scores indicate worse symptoms and a greater impact on quality of life.
  Breakdown: The score is the sum of three items: frequency (0-5), amount (0-6), and interference with everyday life (0-10).

SECONDARY OUTCOMES:
PERFECT scheme | 12 weeks
  This is used to evaluate Pelvic Floor Muscle Function. It evaluates four components: Power, Endurance, Repetitions, and Fast contractions. Higher scores indicate better muscle function
Surface electromyography | 12 weeks
  This is used to evaluate Core and Pelvic Floor Muscle Activation
Urogenital Distress Inventory (UDI-6) | 12 weeks
  This questionnaire assesses the degree of bother associated with specific urogenital symptoms (e.g., frequent urination, leakage).
  Minimum Score: 0
  Maximum Score: 100 (Standardized Scale)
  Interpretation: Higher scores indicate worse quality of life (higher distress).
  Calculation: There are 6 items. Each is rated 0 (Not at all) to 3 (Greatly). The average score of the items is calculated and then multiplied by 33.33 to convert it to a 0-100 scale.
the Incontinence Impact Questionnaire (IIQ-7) | 12 weeks
  This questionnaire measures the impact of urinary incontinence on activities, roles, and emotional health.
  Minimum Score: 0
  Maximum Score: 100 (Standardized Scale)
  Interpretation: Higher scores indicate worse quality of life (greater negative impact).
  Calculation: There are 7 items. Each is rated 0 (Not at all) to 3 (Greatly). Like the UDI-6, the average of the item scores is multiplied by 33.33 to obtain the final 0-100 score.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Çınar, Principal Investigator — Bezmialem.edu.tr
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No